CLINICAL TRIAL: NCT03445988
Title: Comparative Effectiveness of Pain Cognitive Behavioral Therapy and Chronic Pain Self-Management Within the Context of Opioid Reduction: The EMPOWER Study
Brief Title: Cognitive Behavioral Therapy and Chronic Pain Self-Management Within the Context of Opioid Reduction: The EMPOWER Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Beth Darnall, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 44918
Record Dates: First submitted 2018-02-15; First posted 2018-02-26 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain
Keywords: opioid, taper, behavioral treatment for pain, randomized
MeSH Terms: conditions — Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The study manager, site coordinators, and clinicians were unblinded to group assignments, while non-clinical study investigators and statisticians remained blinded throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Taper + Cognitive Behavioral Therapy (Active Comparator): A trained psychologist delivers pain-CBT to individual patients or groups of patients with chronic pain. Group treatment is delivered across 8 weekly sessions that last for 2 hours each. Pain-CBT incorporates interactive discussion, practice of relaxation training, action planning, and home exercises into each session. Pain-CBT is effective for reducing pain intensity, pain catastrophizing, depression and social impacts.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Taper + Chronic Pain Self Management Program (Active Comparator): The CPSMP is similar to pain-CBT in format and content but is peer-led, and is effective across pain conditions (e.g., back pain, arthritis) for improving pain and pain self-efficacy. The CPSMP consists of six weekly 2-hour group sessions in which two peer co-leaders provide patient education about pain, effective self-management, pain impacts, and other symptoms from a highly structured manual. Peers are people with chronic pain who live in the communities in which they teach. For this project, at least one peer facilitator per workshop will have had experience with prescription opioid use. Intervention fidelity is determined by having a trained observer with a checklist attend random workshop sessions. Similar to pain-CBT, CPSMP incorporates interactive discussion, practice of relaxation training, action planning, and home exercises into each session.
  Interventions: Behavioral: Chronic Pain Self Management Program
- Taper Only (no assigned behavioral treatment) (Placebo Comparator): Participants allocated to 'Taper Only' will engage in a physician-guided, patient-centered opioid tapering program without additional behavioral intervention.
  Interventions: Other: Taper Only
- National Observational Study (non-randomized) (No Intervention): The national observational arm of the study (the VALUE study) will enroll participants with chronic pain taking at least 10 MEDD daily. No interventions of any kind will be applied and only self-report survey data will be collected for the year following consent. EMPOWER (randomized trial) and VALUE are two independent studies. Data from the two studies will be analyzed separately.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — A trained psychologist delivers pain-CBT to individual patients or groups of patients with chronic pain. Group treatment is delivered across 8 weekly sessions that last for 2 hours each. Pain-CBT incorporates interactive discussion, practice of relaxation training, action planning, and home exercises into each session. Pain-CBT is effective for reducing pain intensity, pain catastrophizing, depression and social impacts.
  Arms: Taper + Cognitive Behavioral Therapy
Behavioral: Chronic Pain Self Management Program — The CPSMP is similar to pain-CBT in format and content but is peer-led, and is effective across pain conditions (e.g., back pain, arthritis) for improving pain and pain self-efficacy. The CPSMP consists of six weekly 2-hour group sessions in which two peer co-leaders provide patient education about pain, effective self-management, pain impacts, and other symptoms from a highly structured manual. Similar to pain-CBT, CPSMP incorporates interactive discussion, practice of relaxation training, action planning, and home exercises into each session
  Arms: Taper + Chronic Pain Self Management Program
Other: Taper Only — Participants allocated to 'Taper Only' will engage in a physician-guided, patient-centered opioid tapering program without additional behavioral intervention.
  Arms: Taper Only (no assigned behavioral treatment)

SUMMARY:
The proposed study will fill several critical gaps in evidence that are preventing patients and physicians from making informed decisions about their pain care. This project will provide patients taking opioids and physicians with the specific evidence they need to choose the most effective route to pain control, reduced pain interference, opioid reduction, and improved role function, thereby improving patient care.

The aims of this study are to (1) reduce or contain prescription opioid use while maintaining pain control and (2) compare the effectiveness of the Chronic Pain Self-Management Program (CPSMP), Cognitive Behavioral Therapy for chronic pain (pain-CBT), and no behavioral treatment within the context of patient-centered collaborative opioid tapering (Taper Only).

The acronym EMPOWER stands for Effective Management of Pain and Opioid-Free Ways to Enhance Relief.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-cancer pain (≥ 6 months in duration)
* Currently receiving prescription opioids (≥ 10 MEDD) for ≥ 3 months

Exclusion Criteria:

* Unable to provide informed consent
* Unable to participate in group treatments in a meaningful way (e.g., evident cognitive impairment or lack of English fluency)
* Moderate to severe opioid use disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1462 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Darnall, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We partnered with seven study sites that included four outpatient primary care and Veterans health care and three pain clinics in five states (Arizona, California, Colorado, Pennsylvania, and Utah). At all sites, patient recruitment (August 2018-November 2022) was enhanced by using several methods: identifying eligibility in medical records, in-house advertising, external community-based advertising, and use of the CHOIR database at Stanford University.
Pre-assignment Details: EMPOWER (opioid taper study; 3-arm randomized): 53 patients who provided consent did not complete their baseline survey; 562 participants completed their baseline survey and were randomized.
  VALUE (national observational study; non-randomized): 37 individuals who provided consent did not complete their baseline survey; 810 participants completed their baseline survey.
Groups:
- Cognitive Behavioral Therapy for Chronic Pain (Pain-CBT): A trained psychologist delivers pain-CBT to individual patients or groups of patients with chronic pain. Group treatment is delivered across 8 weekly sessions that last for 2 hours each. Pain-CBT incorporates interactive discussion, practice of relaxation training, action planning, and home exercises into each session. Pain-CBT is effective for reducing pain intensity, pain catastrophizing, depression and social impacts.
- Chronic Pain Self Management Program (CPSMP): The CPSMP is similar to pain-CBT in format and content but is peer-led, and is effective across pain conditions (e.g., back pain, arthritis) for improving pain and pain self-efficacy. The CPSMP consists of six weekly 2-hour group sessions in which two peer co-leaders provide patient education about pain, effective self-management, pain impacts, and other symptoms from a highly structured manual. Peers are people with chronic pain who live in the communities in which they teach. For this project, at least one peer facilitator per workshop will have had experience with prescription opioid use. Intervention fidelity is determined by having a trained observer with a checklist attend random workshop sessions. Similar to pain-CBT, CPSMP incorporates interactive discussion, practice of relaxation training, action planning, and home exercises into each session.
- Taper Only (Usual Care): Participants allocated to 'Taper Only' will engage in a physician-guided, patient-centered opioid tapering program without additional behavioral intervention.
- Observational Arm (The VALUE Study): Participants that do not wish to reduce their opioid medications but are otherwise eligible and interested in the research study will be offered participation in the observational arm. The observational arm of the study will not include interventions of any kind and will only collect survey data for the year following consent.
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy for Chronic Pain (Pain-CBT) | Chronic Pain Self Management Program (CPSMP) | Taper Only (Usual Care) | Observational Arm (The VALUE Study)
Started | 203 | 168 | 191 | 810
Completed | 177 | 137 | 159 | 735
Not Completed | 26 | 31 | 32 | 75
Not completed — Lost to Follow-up | 14 | 26 | 27 | 66
Not completed — Withdrawal by Subject | 7 | 4 | 3 | 5
Not completed — Death (unrelated to study) | 5 | 1 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
Groups:
- Observational Arm (the VALUE Study): Participants that do not wish to reduce their opioid medication(s) but are otherwise eligible and interested in the research study will be offered participation in the observational arm. The observational arm of the study will not include interventions of any kind and will only collect survey data for the year following consent. Data from the VALUE study will be analyzed separately from EMPOWER (randomized).
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy for Chronic Pain (Pain-CBT) | Chronic Pain Self Management Program (CPSMP) | Taper Only (Usual Care) | Observational Arm (the VALUE Study) | Total
Number analyzed (Participants) | 203 | 168 | 191 | 810 | 1372
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  years
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 58 (13) | 59 (12) | 56 (13) |  | 58 (13)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 54.5 (10.8) | 54.5 (10.8)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  Participants
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized): Female | 113 | 79 | 104 |  | 296
    EMPOWER Study (randomized): Male | 90 | 89 | 87 |  | 266
    EMPOWER Study (randomized): Unknow or not reported | 0 | 0 | 0 |  | 0
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized): Female |  |  |  | 652 | 652
    VALUE Study (non-randomized): Male |  |  |  | 154 | 154
    VALUE Study (non-randomized): Unknow or not reported |  |  |  | 4 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  Participants
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized): Hispanic or Latino | 24 | 12 | 22 |  | 58
    EMPOWER Study (randomized): Not Hispanic or Latino | 174 | 152 | 159 |  | 485
    EMPOWER Study (randomized): Unknown or Not Reported | 5 | 4 | 10 |  | 19
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized): Hispanic or Latino |  |  |  | 43 | 43
    VALUE Study (non-randomized): Not Hispanic or Latino |  |  |  | 756 | 756
    VALUE Study (non-randomized): Unknown or Not Reported |  |  |  | 11 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  Participants
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized): American Indian or Alaska Native | 0 | 0 | 0 |  | 0
    EMPOWER Study (randomized): Asian | 3 | 4 | 0 |  | 7
    EMPOWER Study (randomized): Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0
    EMPOWER Study (randomized): Black or African American | 9 | 10 | 7 |  | 26
    EMPOWER Study (randomized): White | 154 | 127 | 150 |  | 431
    EMPOWER Study (randomized): More than one race | 14 | 11 | 8 |  | 33
    EMPOWER Study (randomized): Unknown or Not Reported | 23 | 16 | 26 |  | 65
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized): American Indian or Alaska Native |  |  |  | 0 | 0
    VALUE Study (non-randomized): Asian |  |  |  | 4 | 4
    VALUE Study (non-randomized): Native Hawaiian or Other Pacific Islander |  |  |  | 0 | 0
    VALUE Study (non-randomized): Black or African American |  |  |  | 10 | 10
    VALUE Study (non-randomized): White |  |  |  | 718 | 718
    VALUE Study (non-randomized): More than one race |  |  |  | 38 | 38
    VALUE Study (non-randomized): Unknown or Not Reported |  |  |  | 40 | 40
Pain Duration [Count of Participants; unit: Participants] — Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  Participants
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized): 0.5 - 1 year | 1 | 0 | 2 |  | 3
    EMPOWER Study (randomized): 1 - 5 years | 24 | 28 | 32 |  | 84
    EMPOWER Study (randomized): 6 - 10 years | 25 | 26 | 23 |  | 74
    EMPOWER Study (randomized): 10 - 20 years | 76 | 57 | 68 |  | 201
    EMPOWER Study (randomized): > 20 years | 76 | 57 | 66 |  | 199
    EMPOWER Study (randomized): Unknown or not reported | 1 | 0 | 0 |  | 1
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized): 0.5 - 1 year |  |  |  | 7 | 7
    VALUE Study (non-randomized): 1 - 5 years |  |  |  | 48 | 48
    VALUE Study (non-randomized): 6 - 10 years |  |  |  | 145 | 145
    VALUE Study (non-randomized): 10 - 20 years |  |  |  | 301 | 301
    VALUE Study (non-randomized): > 20 years |  |  |  | 302 | 302
    VALUE Study (non-randomized): Unknown or not reported |  |  |  | 7 | 7
Pain Intensity - Average [Mean (Standard Deviation); unit: units on a scale] — Pain intensity was assessed with the Patient Reported Outcomes Measurement Systems (PROMIS) Pain Intensity 1-item scale assessing average pain intensity for the past 7 days (0= "No pain" to 10= "Worst pain imaginable") where a higher score represents a greater degree of pain intensity. Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  units on a scale
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 6.2 (1.9) | 6.2 (1.9) | 6.2 (1.9) |  | 6.2 (1.9)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 6.1 (1.8) | 6.1 (1.8)
Morphine Equivalent Daily Dose (MEDD) [Mean (Standard Deviation); unit: MEDD] — Daily opioid doses were converted to standardized MEDD using the 2016 CDC Guidelines, including the adjusted methadone conversion factor for higher doses. Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  MEDD
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 141.6 (280.0) | 123.4 (263.0) | 109.1 (167.0) |  | 125.1 (242.0)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 116 (194) | 116 (194)
Pain Catastrophizing Scale [Mean (Standard Deviation); unit: score on a scale] — The pain catastrophizing scale (PCS) has 13 items and measures patterns of negative thoughts and emotional responses to pain. The response scale ranges from 0 (not at all) to 4 (all the time); total sum scores range from 0 to 52, with higher scores indicating greater pain catastrophizing tendencies. Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  score on a scale
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 20.8 (11.6) | 22.8 (11.9) | 21.6 (11.5) |  | 21.7 (11.7)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 32.4 (12.0) | 32.4 (12.0)
Brief Pain Inventory (BPI) - Pain Interference [Mean (Standard Deviation); unit: units on a scale] — The BPI assess the level of pain-related interference across the following seven domains: mood, general activity, normal work (inside and outside the home), enjoyment of life, relations with other people, walking ability, and sleep (0=does not interfere, 10=completely interferes). Higher scores signify worse pain interference. The average score (range from 0 to 10) was created by averaging the seven domain scores for each participant. Population: Different measure was used to assess pain interference in the VALUE study. Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  units on a scale
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 5.9 (2.4) | 5.8 (2.3) | 6.1 (2.2) |  | 5.9 (2.3)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
PROMIS - Pain Interference [Mean (Standard Deviation); unit: score on a scale] — A score of 50 is the average for the United States general population with a standard deviation of 10; therefore, a person with a T-score of 40 is one SD below the mean. A higher score indicates greater symptom severity. Population: Different measure was used in the EMPOWER study to assess for pain interference. Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  score on a scale
    EMPOWER Study (randomized): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 68.1 (6.0) | 68.1 (6.0)
Pain Self-Efficacy [Mean (Standard Deviation); unit: units on a scale] — The 2-item Pain Self-Efficacy Questionnaire assessed confidence in functioning in the presence of pain. Responses range from 0 = "Not at all confident" to 6 = "Completely confident" where higher scores represent greater confidence in functioning. Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  units on a scale
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 6.2 (3.6) | 6.6 (3.3) | 6.7 (3.4) |  | 6.5 (3.4)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 5.4 (3.4) | 5.4 (3.4)
PROMIS - Anger [Mean (Standard Deviation); unit: score on a scale] — A score of 50 is the average for the United States general population with a standard deviation of 10; therefore, a person with a T-score of 40 is one SD below the mean. A higher score indicates greater symptom severity. Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  score on a scale
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 49.9 (9.4) | 49.9 (8.9) | 51.3 (9.0) |  | 50.4 (9.1)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 49.3 (9.3) | 49.3 (9.3)
PROMIS - Anxiety [Mean (Standard Deviation); unit: score on a scale] — A score of 50 is the average for the United States general population with a standard deviation of 10; therefore, a person with a T-score of 40 is one SD below the mean. A higher score indicates greater symptom severity. Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  score on a scale
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 54.6 (9.7) | 54.5 (9.5) | 55.9 (9.4) |  | 55.0 (9.6)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 53.0 (9.1) | 53.0 (9.1)
PROMIS - Cognitive Function [Mean (Standard Deviation); unit: score on a scale] — A score of 50 is the average for the United States general population with a standard deviation of 10; therefore, a person with a T-score of 40 is one SD below the mean. A higher score indicates greater symptom severity. Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  score on a scale
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 53.6 (10.4) | 54.4 (9.9) | 55.4 (9.7) |  | 54.5 (10.0)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 53.2 (10.0) | 53.2 (10.0)
PROMIS - Physical Function [Mean (Standard Deviation); unit: score on a scale] — A score of 50 is the average for the United States general population with a standard deviation of 10; therefore, a person with a T-score of 40 is one SD below the mean. A higher score indicates greater symptom severity. Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  score on a scale
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 64.8 (6.5) | 63.9 (6.1) | 64.4 (6.5) |  | 64.4 (6.4)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 65.4 (5.3) | 65.4 (5.3)
PROMIS - Fatigue [Mean (Standard Deviation); unit: score on a scale] — A score of 50 is the average for the United States general population with a standard deviation of 10; therefore, a person with a T-score of 40 is one SD below the mean. A higher score indicates greater symptom severity. Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  score on a scale
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 57.7 (10.0) | 56.8 (9.3) | 58.2 (9.6) |  | 57.6 (9.7)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 60.3 (9.8) | 60.3 (9.8)
PROMIS - Sleep Disturbance [Mean (Standard Deviation); unit: score on a scale] — A score of 50 is the average for the United States general population with a standard deviation of 10; therefore, a person with a T-score of 40 is one SD below the mean. A higher score indicates greater symptom severity. Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  score on a scale
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 57.4 (8.6) | 55.5 (8.8) | 57.4 (8.3) |  | 56.8 (8.6)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 57.2 (8.5) | 57.2 (8.5)
PROMIS - Social Isolation [Mean (Standard Deviation); unit: score on a scale] — A score of 50 is the average for the United States general population with a standard deviation of 10; therefore, a person with a T-score of 40 is one SD below the mean. A higher score indicates greater symptom severity. Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  score on a scale
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 47.4 (9.5) | 48.8 (9.3) | 48.7 (9.7) |  | 48.3 (9.5)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 48.9 (9.3) | 48.9 (9.3)
PROMIS - Satisfaction with Social Roles & Activities [Mean (Standard Deviation); unit: score on a scale] — A score of 50 is the average for the United States general population with a standard deviation of 10; therefore, a person with a T-score of 40 is one SD below the mean. A higher score indicates greater symptom severity. Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  score on a scale
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 59.8 (8.1) | 58.5 (7.5) | 60.1 (7.7) |  | 59.5 (7.8)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 60.4 (7.8) | 60.4 (7.8)
PROMIS - Depression [Mean (Standard Deviation); unit: score on a scale] — A score of 50 is the average for the United States general population with a standard deviation of 10; therefore, a person with a T-score of 40 is one SD below the mean. A higher score indicates greater symptom severity. Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  score on a scale
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 54.8 (8.9) | 55.3 (8.0) | 55.9 (8.8) |  | 55.3 (8.6)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 54.6 (8.7) | 54.6 (8.7)
Alcohol Use Disorders Identification Test (AUDIT) [Mean (Standard Deviation); unit: score on a scale] — A total score (range: 0 to 40) is calculated by adding the points for each item which have a response scale of either 0 to 2 or 0 to 4. A score of 8 or more is associated with harmful or hazardous drinking, a score of 13 or more in women, and 15 or more in men, is likely to indicate alcohol dependence. Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  score on a scale
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 0.9 (2.3) | 1.3 (2.4) | 0.9 (2.0) |  | 1.0 (2.2)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 1.4 (2.1) | 1.4 (2.1)
Drug Abuse Screen Test (DAST) [Mean (Standard Deviation); unit: score on a scale] — A total score (range: 0-10) is calculated by adding the points for each item of the ten items. Score of 0: No problems reported; 1-2: Low level; 3-5: Moderate level; 6-8: Substantial level; 9-10: Severe level. Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately.
  score on a scale
    EMPOWER Study (randomized): number analyzed (Participants) | 203 | 168 | 191 | 0 | 562
    EMPOWER Study (randomized) | 0.6 (1.2) | 0.6 (1.3) | 0.5 (1.2) |  | 0.6 (1.2)
    VALUE Study (non-randomized): number analyzed (Participants) | 0 | 0 | 0 | 810 | 810
    VALUE Study (non-randomized) |  |  |  | 2.1 (1.4) | 2.1 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Tapering Success
Description: Opioid tapering success was defined as either: 50% reduction in opioid dose (change in MEDD baseline to 12 months) and no significantly increased pain (≤ 1 point increase in PROMIS pain intensity score from baseline to 12 months), or; no opioid dose increase (baseline MEDD to 12 months) and significant pain relief (≥ 2 points decrease in PROMIS pain intensity score). Pain intensity score: Patient self-reported pain intensity on 11 point (0-10) numerical rating scale where a lower score means more pain relief. MEDD: Morphine Equivalent Daily Dose. PROMIS: Patient-Reported Outcomes Measurement Information System.
Time Frame: Baseline and 12 months
Population: Data from the two studies (EMPOWER and VALUE) were analyzed separately. VALUE study did not have opioid tapering success as an outcome given that the study was observational (there was no opioid tapering implemented as part of the study); therefore, participants in the VALUE study were not assessed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioral Therapy for Chronic Pain (Pain-CBT) | Chronic Pain Self Management Program (CPSMP) | Taper Only (Usual Care) | Observational Arm (The VALUE Study)
Number analyzed (Participants) | 177 | 137 | 159 | 0
Participants | 86 | 61 | 81 | 0

ADVERSE EVENTS:
Time Frame: Baseline, Weekly, Month 6, Monthly, and Month 12.
Arm/Group | Cognitive Behavioral Therapy for Chronic Pain (Pain-CBT) | Chronic Pain Self Management Program (CPSMP) | Taper Only (Usual Care) | Observational Arm (the VALUE Study)
All-Cause Mortality (participants affected / at risk) | 5/203 | 1/168 | 2/191 | 4/810
Serious Adverse Events (participants affected / at risk) | 9/203 | 7/168 | 8/191 | 0/810
Other Adverse Events (participants affected / at risk) | 162/203 | 140/168 | 159/191 | 0/810
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cognitive Behavioral Therapy for Chronic Pain (Pain-CBT) (N=203) | Chronic Pain Self Management Program (CPSMP) (N=168) | Taper Only (Usual Care) (N=191) | Observational Arm (the VALUE Study) (N=810)
Car accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1 | 0
Surgery - elective (Surgical and medical procedures) | 2 | 1 | 0 | 0
Differential diagnosis (General disorders) | 0 | 0 | 1 | 0
Cardiac issue (Cardiac disorders) | 0 | 0 | 1 | 0
(General disorders) | 1 | 0 | 1 | 0
Parkinson's disease (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Progressive chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
cerebrovascular accident (stroke) (Vascular disorders) | 0 | 0 | 3 | 0
Decompensated heart failure (Cardiac disorders) | 1 | 0 | 0 | 0
Alcohol use complications (General disorders) | 1 | 0 | 0 | 0
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Failing kidneys (Renal and urinary disorders) | 1 | 0 | 0 | 0
Toe amputation (Surgical and medical procedures) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cognitive Behavioral Therapy for Chronic Pain (Pain-CBT) (N=203) | Chronic Pain Self Management Program (CPSMP) (N=168) | Taper Only (Usual Care) (N=191) | Observational Arm (the VALUE Study) (N=810)
Emergency room visit (General disorders) | 31 | 20 | 33 | 0
Medical history - chronic pain (Nervous system disorders) | 33 | 61 | 26 | 0
New medical issue (General disorders) | 68 | 35 | 44 | 0
Urgent care visit (General disorders) | 4 | 4 | 7 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Subjective Opiate Withdrawal Scale (SOWS) (General disorders) | 26 | 20 | 48 | 0

LIMITATIONS AND CAVEATS:
COVID-related challenges resulted in a smaller sample size than was planned. Results may not generalize to those with less education or racial/ethnic diversity. Results do not generalize to patients with moderate to severe opioid use disorder, and are limited to our specific voluntary patient-centered tapering methods. The supportive and real-time responsive communication platform used across all study arms may have biased results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03445988/Prot_SAP_ICF_000.pdf